CLINICAL TRIAL: NCT02905045
Title: Effect of Oral Ketoprofen on Hysterosalpingography Pain: A Randomized Controlled Trial
Brief Title: Efficacy of Ketoprofen Before Hysterosalpingography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KETOHSG
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pain Relief
MeSH Terms: interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketoprofen (Active Comparator): women will take one tablet 150 mg one hour before the procedure
  Interventions: Drug: Ketoprofen
- Placebo (Placebo Comparator): women will take one tablet placebo one hour before the procedure
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ketoprofen
  Other Names: bi profenid
  Arms: Ketoprofen
Drug: placebo
  Arms: Placebo

SUMMARY:
hysterosalpingography can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the cannula; and injection of the dye

ELIGIBILITY:
Inclusion Criteria:

* any patient came for Hysterosalpingography

Exclusion Criteria:

* any patient has contraindication to Hysterosalpingography

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Mean pain score during the procedure | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided